CLINICAL TRIAL: NCT04501419
Title: Tablet-based Mobile Health Ultrasound for Point-of-care Breast Cancer Diagnosis in Nigeria
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Obafemi Awolowo University Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ERC/2019/10/05; 18-114 (Other: Memorial Sloan Kettering Cancer Center)
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trained radiologists (Experimental): Trainers will successfully train Nigerian radiologists
  Interventions: Other: Ultrasound-guided breast biopsy training program
- Patients with a suspicious breast mass (Experimental): Women that present to the hospital with a suspicious breast mass
  Interventions: Procedure: US-guided breast biopsy

INTERVENTIONS:
Procedure: US-guided breast biopsy — During this study, women with undergo an US-guided breast biopsy by a radiologist instead of what is typically performed in Nigerian hospitals, which is either a blind biopsy or surgical excision. US-guided breast biopsy is the standard of care in the United States of America because the accuracy is better than blind biopsy and equal to surgical excision.
  Arms: Patients with a suspicious breast mass
Other: Ultrasound-guided breast biopsy training program — This program, developed by experts in Nigeria and the United States of America, certifies that they have the skills required to safely perform these biopsies on patients
  Arms: Trained radiologists

SUMMARY:
The purpose of this study is to train Nigerian radiologists to perform ultrasound-guided breast biopsies on women that present to the hospital with a suspicious breast mass. Before performing biopsies on patients, the Nigerian radiologists will have already successfully completed a competency-based mobile health ultrasound-guided breast biopsy-training program. This program, developed by experts in Nigeria and the United States of America, certifies that they have the skills required to safely perform these biopsies on patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older female
* Breast ultrasound demonstrating a solid mass that is suspicious for cancer, which would typically undergo either a blind biopsy or surgical excision at the Nigerian hospital where the patient is seeking diagnosis.

Exclusion Criteria:

* Participants unwilling to sign consent
* Participants under the age of 18.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Enrollment: 600 (Estimated)
Dates: Start 2019-10-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of US-guided breast biopsy in Nigeria compared to reference standard surgical excision | 12 months
  US-guided breast biopsies accuracy measurements will be reported using surgical pathology as the reference standard. Specifically we will report accuracy, positive predictive value, negative predictive value, sensitivity and specificity.

SECONDARY OUTCOMES:
Complication rates from US-guided breast biopsy compared to reference values reported in the literature. | 12 months
  To determine if the complication rate of US-guided breast biopsies performed by the trained Nigerian radiologists is equivalent to reference values reported in the literature.

CONTACTS AND LOCATIONS:
Overall Officials: Adeleye Omisore, MD, Principal Investigator — Obafemi Awolowo University Teaching Hospitals
Locations (1):
- Obafemi Awolowo University Teaching Hospitals Complex (OAUTHC), Ile-Ife, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Omisore AD, Egberongbe AA, Pace LE, Raza S, Akinola RA, Obajimi MO, Sevilimedu V, Bryce Y, Mango VL, Alatise OI, Kingham TP, Morris EA, Sutton EJ. A Competency-Based Ultrasound-Guided Breast Biopsy Training Program for Radiologists From Low-and-Middle-Income Countries that Leverages Mobile Health Technology (NCT04501419): A Study Protocol. Cancer Control. 2025 Jan-Dec;32:10732748251334435. doi: 10.1177/10732748251334435. Epub 2025 Apr 18. PMID 40250340